CLINICAL TRIAL: NCT02906449
Title: Investigating the Physiological, Cognitive, and Psychological Effects of a Cognitive-Based Intervention
Acronym: IPCPE-Mind
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brock University (Other)
Responsible Party: Principal Investigator, Dawn Good, Principal Investigator, Brock University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DGBrockU
Record Dates: First submitted 2016-09-15; First posted 2016-09-20 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Brain Concussion, Post-Concussion Syndrome
Keywords: concussion, mild head injury, mindfulness
MeSH Terms: conditions — Brain Concussion; Post-Concussion Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness Training (Experimental): Daily Mindfulness Training - both in-class lectures (weekly) and self-study (daily) over 3 weeks
  Interventions: Behavioral: Meditation Technique
- Relaxation Meditation Training (Active Comparator): Daily Relaxation Meditation Training - both in-class lectures (weekly) and self-study (daily) over 3 weeks
  Interventions: Behavioral: Meditation Technique

INTERVENTIONS:
Behavioral: Meditation Technique — Alertness training or relaxation training

SUMMARY:
The primary purpose of this study is to investigate the effectiveness of a brief mindfulness-based intervention for targeting chronic physiological underarousal and post-concussive symptoms following a mild head injury (MHI), as self-reported by undergraduate university students. For the purposes of this study, MHI is defined (and identified) through our demographic questionnaire as a traumatic-based injury to the head - "Have you ever hit your head with a force sufficient to alter your state of consciousness" (consistent with the Kay et al., 1993 criteria/definition; American Congress of Rehabilitation Medicine - ACRM). The investigators exclude congenital or genetic injuries.

DETAILED DESCRIPTION:
Seventy subjects, aged 17 to 30 years old, from Brock University will be recruited to participate in the study. The ability to speak and write in English is a requirement. University students will be invited to participate in the study in a series of individual and group testing/training sessions (n ≤ 15) on five separate occasions (two testing sessions and three training sessions). The testing/training sessions will be on average, one week apart (depending on the availability of the participants). Participants will be invited to review the consent form prior to the first testing session via having it e-mailed to them once recruited. At this time, a discussion about the student's potential allergies and sensitivities will take place during the review of 'Potential Risks'. Participants will be given two copies of the written consent form to be completed (one copy is given to the participant and the other copy is for the researcher). Subjects will be advised that alternate arrangements can be made if they prefer 'same sex' researchers. All participants will be administered the same protocol and questionnaire order. These tests are well-researched and their standard administration times will be applied.

During the first session (pre-test), participants will be greeted individually for the session in a lab setting in the Jack and Nora Walker Lifespan Development Centre testing facilities at Brock University. The consent form will be read aloud to the participants by the researcher for clarification, and participants will be invited to ask any questions at that time or any time throughout the study. Participants will then undergo a 3-minute physiological recording and complete two performance-based neuropsychological measures: the Trail Making Test (TMT) to measure cognitive flexibility and the Colour-Word Interference Test to measure attention.

For the physiological measures, subjects will be introduced to the Polygraph Professional (2008) equipment which measures heart rate, electrodermal activity (EDA), respiration and blood pressure. Silver-silver chloride pads will be used to collect EDA, and will be placed on the index and fourth fingers on the participant's non-dominant hand. Electrodermal activation (EDA) responses are measured in terms of amplitude (i.e., the height of the electrodermal response measured in microsiemens [µS]). A pulse oximeter will be placed on the middle finger of the participant's non-dominant hand to measure HR. Respiration will be recorded via two pneumatic chest bands - the upper will be placed around the chest and the lower, around the abdomen and over their clothing. Blood pressure will be measured via a blood pressure cuff that will be placed on the brachial artery/upper portion of the individual's left arm. All core equipment is cleansed with alcohol swabs after use; the researcher will provide the participant with antibacterial lotion prior to application of electrodes; electrodes will be replaced as needed. The sanitary procedures will be explained to the subject and implemented (e.g., experimenter's use of gloves, and use of cleansed and disinfected equipment using alcohol, etc.).

In addition, the participant will be asked to complete a self-report rating of his/her arousal level before physiological activity is recorded (as used in, for example, Baker and Good [2014], participants are shown a scale (from 1 to 10) on a laminated sheet and asked to provide a self-report rating of their current arousal state (1 - e.g., very relaxed to 10 - e.g., very stressed). Subjects will be seated and will be given time to rest prior to, and during, the recordings. Participants will be asked to remain still in a relaxed and comfortable position (to reduce physical movement) while a recording is taken for a 3- minute period. All physiological data recorded will be coded alphanumerically without personal identifiers.

Following the physiological recordings, the Trail Making Test will be administered, during which the subjects are asked to connect a series of numbered and lettered dots according to a specific set of rules. Subsequently, the Colour-Word Interference Test will be administered, during which subjects are asked to read aloud the colour of ink that various colour words are printed in. All neurocognitive tests will be administered under time constraints as dictated by testing protocol. The participant will then be accompanied to a separate (nearby) room to complete a selection of self-report questionnaires in a group testing environment (i.e., with up to 14 other participants). Note: the BDI-II will be scored immediately after the student has completed testing (i.e., immediately after they leave the testing session).

During this group testing session, participants will be asked to complete a selection of untimed, self-paced self-report questionnaires that measure the following: psychopathology - e.g., depressive and anxiety symptoms (Beck Depression Inventory [BDI], Beck Anxiety Inventory [BAI]); executive functioning (Behavior Rating Inventory of Executive Function - Adult [BRIEF-A]); trait mindfulness (Five Facet Mindfulness Questionnaire [FFMQ]), personality characteristics (HEXACO Personality Inventory - Revised [HEXACO-PI-R]) and lastly demographics (Everyday Living Questionnaire), which includes a measure of post-concussive symptoms (Post-Concussion Symptom Scale [PCS]). The first session is expected to take approximately 1.5 hours to complete in total.

Following the completion of the first testing session, participants will be instructed to sign-up for a cognitive training session, which will take place within one week following the pre-test session. Participants will be randomly assigned to either a mindfulness training session (experimental group; n = 35) or a relaxation training session (control group; n = 35).

Both the mindfulness training group and the relaxation training group will meet for approximately 30 minutes each week, across three separate training sessions. Participants will be greeted as a group for the session in a lab setting in the Jack and Nora Walker Lifespan Development Centre testing facilities at Brock University. Participants in the mindfulness training group will partake in an interactive training session, which will involve learning core mindfulness-related concepts, as well as engaging in progressively advanced mindfulness exercises. Note: For exercises involving the consumption of food products, participants will be notified in advance (and immediately before the exercises) of the food products that will be involved in the exercise. Participants will be cautioned to take into consideration any food allergies and/or dietary restrictions they may have - precautions will be taken such that the risk of food allergies is minimized (e.g., selecting foods that are nut-free). Following the formal mindfulness sessions, participants will be instructed to complete daily "homework" exercises (for approximately 5 minutes per day), which will be accessible as handouts and audio recordings on a Brock University Sakai site. Participants will be asked to complete an online questionnaire (taking approximately one minute to complete) each day to record details regarding their daily mindfulness practice.

The procedure for the relaxation training sessions will be similar to the mindfulness sessions. Participants in the relaxation training group will partake in an interactive training session, which will involve learning about the link between stress and cognition, as well as engaging in progressively advanced relaxation techniques focused on reducing anxiety or stress prior to cognitively-demanding tasks. Following the formal relaxation sessions, participants will be instructed to complete daily "homework" exercises (for approximately 5 minutes per day), which will be accessible as handouts and audio recordings on a Brock University Sakai site. Participants will be asked to complete an online questionnaire (taking approximately one minute to complete) each day to record details regarding their daily relaxation practice.

At the end of every training session (for the mindfulness group and control group), participants will be asked to complete a short self-report questionnaire, measuring state mindfulness (i.e., the Toronto Mindfulness Scale [TMS]).

During the final session (post-test), participants will be greeted individually for the session in a lab setting in the Jack and Nora Walker Lifespan Development Centre testing facilities at Brock University. The post-test session will follow the same procedure as the pre-test session (as described earlier). Participants will complete the same physiological, neuropsychological, and self-report measures as described in the pre-test session, with two exceptions: (1) a shorter version of the Everyday Living Questionnaire (and attached Post-Concussion Symptom Scale) will be used to assess changes in post-concussive symptoms since the first testing session. As well, athletic, educational, familial, and pre-test medical history information will not be reassessed. The post-test session will take approximately 1.5 hours to complete.

Upon completion of the study (at the end of the post-test session), participants will be debriefed as to the nature and purpose of the study, and thanked for their participation. Overall, participation in the study will not exceed 6 hours. Included in the debriefing form is counselling contact information for Brock University Counselling Services should any negative emotions surface as a result of participation in the study. Participants will also receive contact information for the principal investigator/faculty supervisor, principal and co-student investigators. Finally, participants will be thanked for their time and participation, and will be invited to review the results of the study at its completion (by August 2017).

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled in University

Exclusion Criteria:

* Individuals with food allergies associated with chocolate
* Individuals with skin sensitivities (e.g., with respect to electrode conductive gel)

Ages: 17 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Five Facet Mindfulness Questionnaire | 5 weeks from the beginning of the study
  The FFMQ is a trait measure of mindfulness (end point minus baseline)
Beck Depression Inventory - 2 | 5 weeks from the beginning of the study
  Measures the intensity of depressive symptoms (end point minus baseline)
Beck Anxiety Inventory | 5 weeks from the beginning of the study
  Measures the intensity of anxiety symptoms (end point minus baseline)
Autonomic Presentation | 5 weeks from the beginning of the study
  Sympathetic Nervous System measures - EDA, heart rate, blood pressure
Toronto Mindfulness Scale | 5 weeks from the beginning of the study
  Measure of state mindfulness (end point minus baseline)

SECONDARY OUTCOMES:
Trail Making Test | 5 weeks from the beginning of the study
  An index of non-verbal cognitive flexibility
Color-Word Interference Test | 5 weeks from the beginning of the study
  Measures attention and inhibitory control
Behaviour Rating Inventory of Executive Function - Adult version | 5 weeks from the beginning of the study
  Measures self-report deficits in executive functioning
HEXACO Personality Inventory - Revised | 5 weeks from the beginning of the study
  Assesses the six major dimensions of personality

CONTACTS AND LOCATIONS:
Overall Officials: Dawn E Good, PhD, CPsych, Principal Investigator — Brock University

IPD SHARING:
Plan to Share IPD: No
Only congregate/group statistical data will be shared and published

REFERENCES:
- [Background] Bonow, R.O., Mann, D.L., Zipes, D.P., & Libby, P. (2012). Braunwald's Heart Disease: A Textbook of Cardiovascular Medicine. 9th ed. New York: Saunders.
- [Result] Bishop, S. R., Lau, M., Shapiro, S., Carlson, L., Anderson, N. D., Carmody, J., ... & Devins, G. (2004). Mindfulness: A proposed operational definition. Clinical psychology: Science and practice, 11(3), 230-241.
- [Result] Baker JM, Good DE. Physiological emotional under-arousal in individuals with mild head injury. Brain Inj. 2014;28(1):51-65. doi: 10.3109/02699052.2013.857787. PMID 24328800
- [Result] Lau MA, Bishop SR, Segal ZV, Buis T, Anderson ND, Carlson L, Shapiro S, Carmody J, Abbey S, Devins G. The Toronto Mindfulness Scale: development and validation. J Clin Psychol. 2006 Dec;62(12):1445-67. doi: 10.1002/jclp.20326. PMID 17019673
- [Result] Baer RA, Smith GT, Hopkins J, Krietemeyer J, Toney L. Using self-report assessment methods to explore facets of mindfulness. Assessment. 2006 Mar;13(1):27-45. doi: 10.1177/1073191105283504. PMID 16443717
- [Result] Short, M. M., Mazmanian, D., Oinonen, K., & Mushquash, C. J. (2016). Executive function and self-regulation mediate dispositional mindfulness and well-being. Personality and Individual Differences, 93, 97-103. doi:10.1016/j.paid.2015.08.007
- [Result] Brown KW, Ryan RM. The benefits of being present: mindfulness and its role in psychological well-being. J Pers Soc Psychol. 2003 Apr;84(4):822-48. doi: 10.1037/0022-3514.84.4.822. PMID 12703651